CLINICAL TRIAL: NCT07160504
Title: Is There an Effect of Local Vaginal Estrogen Treatment on the Hemostatic Parameters in Postmenopausal Women?
Brief Title: Vaginal Estrogen Treatment and Effect on Hemostatic Parameters in Postmenopausal Women
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-519539-41-00; 2024-519539-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-13; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Vagina Atrophy
Keywords: Postmenopausal; Hemostasis; Venous thromboembolic event

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaginal estrogen treatment (Other)
  Interventions: Drug: Vaginal estradiol tablets

INTERVENTIONS:
Drug: Vaginal estradiol tablets — Vaginal estrogen tablets 10 µg at least 3 times a week (on indication, prescribed at the outpatient clinic).

SUMMARY:
This study investigates whether vaginal estrogen treatment has an effect on hemostatic parameters in postmenopausal women. Blood samples are collected before and after 3 months treatment to assess changes in hemostasis.

DETAILED DESCRIPTION:
This prospective cohort study includes 90 postmenopausal women aged ≥ 50, having vaginal atrophy symptoms and indication for treatment with vaginal estrogen tablets 10 µg at least 3 times a week for 3 months. Participants are divided into 2 study populations. Study population 1: 45 without a history of venous thromboembolic event and study population 2: 45 with a history of venous thromboembolic event.

Participation will involve 2 visits:

* First visit: prior the initiation of treatment an interview is carried out to assess inclusion criteria and information on demographics followed by blood sampling.
* Second visit: follow-up blood sampling after three months treatment. Hemostatic parameters will be assessed, comparing the blood samples at baseline with the follow-up blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged ≥ 50
* Symptomatic vaginal atrophy
* Indication for standard treatment with vaginal estrogen tablets 10 µg at least three times a week
* Study population 1: without a history of venous thromboembolic event
* Study population 2: with a history of venous thromboembolic event

Exclusion Criteria:

* Unable to give written informed consent
* Does not speak Danish
* Current cancer treatment
* Current treatment with blood thinning medication (except plateletinhibitor)
* Current treatment with local or systematic estrogen
* Systemic inflammatory disease, liver disease or kidney disease

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Endogenous thrombin potential (ETP) | 0 months, 3 months
  nmol/l x min
Endogenous trombin lag time (LT) | 0 months, 3 months
  min
Endogenous trombin peak height | 0 months, 3 months
  nmol/l
Factor VIII (FVIII) | 0 months, 3 months
  Percentage
Antithrombin | 0 months, 3 months
  Percentage
Protein S | 0 months, 3 months
  Percentage
Protein C | 0 months, 3 months
  Percentage
D-dimer | 0 months, 3 months
  ng/mL
CRP | 0 months, 3 months
  mg/l
Fibrinogen | 0 months, 3 months
  g/l
Tissue-type plaminogen activator (t-PA) | 0 months, 3 months
  ng/mL
Plasminogen activator inhibitor type 1 (PAI-1) | 0 months, 3 months
  ng/mL
Faktor XII (FXII) | 0 months, 3 months
  μg/mL
Prekallikrein (PK) | 0 months, 3 months
  μg/mL
H-Kininogen (HK) | 0 months, 3 months
  Percentage
Cleaved H-Kininogen (cHK) | 0 months, 3 months
  μg/mL
C1-esterase inhibitor (C1-inh) | 0 months, 3 months
  g/L
Endogenous kallikrein potential (EKP) | 0 months, 3 months
  nmol/L x min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Aarhus University Hospital, Denmark, Aarhus N, Denmark